CLINICAL TRIAL: NCT01296191
Title: Aqueous Absorption and Pharmacokinetics of Besivance Versus VIGAMOX in Patients Undergoing Phacoemulsification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frank A. Bucci, Jr., M.D. (Other)
Responsible Party: Sponsor-Investigator, Frank A. Bucci, Jr., M.D., Principal Investigator, Bucci Laser Vision Institute
Organization: Bucci Laser Vision Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-BV-A
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — Moxifloxacin; besifloxacin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIGAMOX (Active Comparator): Subjects undergoing cataract surgery, randomized to the VIGAMOX group Generic name is moxifloxacin eye drops, drops to be used 1 drop 4 times daily for 3 days prior to surgery and 1 drop on day of surgery.
  Interventions: Drug: Moxifloxacin
- Besivance (Active Comparator): Subjects scheduled for cataract surgery, randomized to the Besivance group Generic name is besifloxacin eye drops, drops to be used 1 drop 4 times daily for 3 days prior to surgery and 1 drop on day of surgery.
  Interventions: Drug: besifloxacin

INTERVENTIONS:
Drug: Moxifloxacin — One drop 4 times daily for 3 days and one drop the day of sample collection
  Other Names: Vigamox
  Arms: VIGAMOX
Drug: besifloxacin — One drop 4 times daily for 3 days and one drop on day of sample collection
  Other Names: Besivance
  Arms: Besivance

SUMMARY:
The purpose of this study is to compare drug concentrations in aqueous humor following ocular instillation of Besivance and VIGAMOX in subjects undergoing cataract surgery.

DETAILED DESCRIPTION:
The objective of this study is to compare drug concentrations in aqueous humor following ocular instillation of Besivance or VIGAMOX in subjects undergoing cataract surgery. The hypothesis of the study is that the aggregate aqueous absorption of Besivance over a six hour period is greater than VIGAMOX because of unique properties of Besivance which promote increased contact time of this antibiotic with the ocular surface.

Subjects with scheduled cataract surgery will be screened during their pre-operative visit. Eligible subjects will be randomized to treatment with Besivance or VIGAMOX. Subjects will self-administer 1 drop of study drug into the operative eye 4 times a day for 3 days prior to surgery.Subjects will have one final drop of study medication on the day of surgery.Immediately prior to beginning the cataract surgery, a sample of aqueous humor will be collected by paracentesis.Concentration of Besivance and VIGAMOX in the aqueous humor will be determined by an independent laboratory using standardized high pressure liquid chromatography and mass spectrometry assays. Pharmacokinetic parameters determined from the aqueous humor concentration-time data will minimally include the area under the curve and the maximum concentration.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 18 years of age or older.
* Physically capable of instilling eye drop or have an appropriate person available to assist in administration of eye drops 4 times a day.
* Scheduled for phacoemulsification with intraocular lens (IOL) implantation for the treatment of cataract.
* Meet the American Society of Anesthesiology (ASA) physical status I, II, or III and be medically cleared for surgery.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Known allergy or contraindication to the test article(s) or their components.
* Presence of any abnormality or significant illness in the eye that in the investigator's opinion could affect the subject's health or the study parameters.
* Presence of an active ocular infection (bacterial, viral or fungal), or positive history of ocular herpetic infection.
* History of any significant illness that could be expected to interfere with the study parameters. Any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study.
* Use of disallowed therapies (systemic or topical):

  * Fluoroquinolone anti-infective agents (systemic or topical) within 1 week of Visit 1 or anytime after Visit 1 for the duration of the study.
* Use of contact lenses for one week prior to the study and for the duration of the study.
* Received an experimental drug or used an experimental medical device within 10 days before the planned start of treatment.
* Breast-feeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank A. Bucci, Jr., MD, Principal Investigator — Bucci Laser Vision Institute
Locations (1):
- Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- VIGAMOX: Subjects undergoing cataract surgery, randomized to the VIGAMOX group
- Besivance: Subjects scheduled for cataract surgery, randomized to the Besivance group
Period: Overall Study
Arm/Group | VIGAMOX | Besivance
Started | 60 | 60
Completed | 57 | 59
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIGAMOX | Besivance | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 51 | 48 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 28 | 63
  Male | 25 | 32 | 57

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics in Aqueous Humor Samples.
Description: Concentration of Besivance and VIGAMOX in the aqueous humor will be determined by an independent laboratory using standardized high-pressure liquid chromatography and mass spectrometry assays. Pharmacokinetic parameters determined from the aqueous humor concentration will minimally include the area under the curve and the maximum concentration.
Time Frame: Measured after 3 days of drug instillation
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | VIGAMOX | Besivance
Number analyzed (Participants) | 57 | 59
ng/ml | 443.07 (232.285) | 56.4525 (39.6325)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the study medications until the aqueous collection. This time period is 4 days.
Arm/Group | VIGAMOX | Besivance
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes